CLINICAL TRIAL: NCT07179393
Title: Evaluating the Efficacy of a Ladies Gaelic Football-Specific Injury Prevention Programme: A Cluster Randomised Trial
Brief Title: Evaluating the Efficacy of a Ladies Gaelic Football-Specific Injury Prevention Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin City University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DCUREC/2025/056
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Injury; Physical Performances
Keywords: Sports Injury Prevention; Community Sport; Ladies Gaelic Football; Injury Prevention Programme
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Cluster Randomised Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Those in the Control Group continue with their regular training/injury prevention practices during the intervention period.
- Intervention Group (Experimental): Those in the Intervention Group perform the injury prevention programme twice weekly as part of their regular training sessions.
  Interventions: Behavioral: Ladies Gaelic Football-Specific Injury Prevention Programme

INTERVENTIONS:
Behavioral: Ladies Gaelic Football-Specific Injury Prevention Programme — This intervention is an injury prevention programme designed with input from Ladies Gaelic football stakeholders (players and coaches) as well as experienced athletic therapy and physiotherapy practitioners and academics from the disciplines of injury prevention and coaching science.
  Arms: Intervention Group

SUMMARY:
The aim of this research is to evaluate the impact of an injury prevention programme on injury risk factors and performance outcomes in Ladies Gaelic Football players. This injury prevention programme was designed with input from Ladies Gaelic football stakeholders and experts and this study will determine if this programme reduces injury risk and improves physical performance over time. Participants will complete physical performance tests before and after the intervention, which consists of incorporating the injury prevention programme into regular team training sessions for 12 weeks. The study will also integrate a qualitative component to assess player's perceptions of the programme and their willingness to implement it.

ELIGIBILITY:
Inclusion Criteria:

* Current Ladies Gaelic Football player competing at adult or minor level from teams consenting to participate in the trial

Exclusion Criteria:

* Players with a current injury preventing full training participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Y-Balance Composite Score | 12 weeks
  Change from pre-testing to post-testing in Ladies Gaelic Football players Y-Balance Composite Score. The Y-Balance Composite Score is a single percentage value from the Y-Balance Test indicating overall stability. Lower scores suggest greater injury risk and higher composite scores suggest less injury risk.
Change in 20 Metre Sprint Time | 12 weeks
  Change in Ladies Gaelic Football players' 20 metre sprint times from pre-testing to post-testing. Lower time is better.
Change in 505 Agility Test Time | 12 weeks
  Change in Ladies Gaelic Football players' 505 Agility Test Time from pre-testing to post-testing. Lower time is better.
Change in Landing Error Scoring System Score | 12 weeks
  Change in Ladies Gaelic Football players' Landing Error Scoring System scores from pre-testing to post-testing. Lower score is better. The minimum possible score is 0 (indicating excellent, low-risk performance), and the maximum possible score is 19 (indicating poor, high-risk performance).
Change in Isometric Hamstring Strength (Maximal Force) | 12 weeks
  Change in Ladies Gaelic Football Isometric Hamstring Strength (Maximal Force) from pre-testing to post-testing as measured by the VALD ForceFrame. Greater Newtons of force is better.
Change in Power Output (measured via a Countermovement Jump) | 12 weeks
  Change in Ladies Gaelic Football players' Power Output (measured via a Countermovement Jump) as measured by the VALD ForceDecks. Greater power output (Watts) is better.

SECONDARY OUTCOMES:
Number of sports-related injuries suffered during the intervention period relative to match hours and training hours (injury incidence) | 12 weeks
  Difference between the control group and intervention group in terms of the number of sports-related injuries suffered during the intervention period relative to match hours and training hours completed by each group
Player/Coach perceptions of the programme and willingness to implement it | 12 weeks
  Interview/Focus groups following the intervention period will assess how players and coaches in the intervention group perceive the injury prevention programme and their willingness to implement it in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- Dublin City University, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided